CLINICAL TRIAL: NCT04501991
Title: Determining the Impact of COVID-19 Lockdown on Metabolic Control in Individuals With Type 2 Diabetes
Brief Title: Short-term Impact of COVID-19 Lockdown on Metabolic Control of Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Anna Solini, Associate Professor, University of Pisa
Other Study IDs: AS0007
Record Dates: First submitted 2020-08-05; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Type 2 Diabetes; Metabolic Control
Keywords: T2D; Sars-Cov-2; COVID-19 lockdown; metabolic control; sedentary
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Type 2 Diabetes: Patients with type 2 diabetes and a scheduled visit during the lockdown for COVID-19
  Interventions: Other: antidiabetic treatment

INTERVENTIONS:
Other: antidiabetic treatment — Every kind of antidiabetic treatment, oral or injective, were considered including patients treated only with diet

SUMMARY:
The strict rules applied in Italy during the recent COVID-19 pandemic, with the prohibition to attend any regular outdoor activity, are likely to influence the degree of metabolic control of patients with type 2 diabetes. The aim of this observational, prospective, single centre study was to evaluate the immediate impact of the lockdown rules on the metabolic profile of a cohort of patients with type 2 diabetes.

DETAILED DESCRIPTION:
All the patients with type 2 diabetes who were previously scheduled for a follow-up visit in our outpatient diabetes clinic during the lockdown for COVID-19 (March 9, 2020-May 04, 2020) were contacted by phone. Patients who accepted to take part of the study received a medical prescription for routine analysis via email. They were asked to perform blood drawing one week after the end of the lockdown period and transmitted us the results.

We then compared the metabolic profile tested one week after the end of the lockdown with the last value and the mean of the last three determinations performed before the pandemic emergency.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* at least two previous clinical records in the last two years

Exclusion Criteria:

* age >85 years
* first access to the outpatient clinic
* type 1 diabetes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients with type 2 diabetes, regularly referring (with at least two previous clinical records in the last two years) to the outpatient diabetes clinic of Internal Medicine section, University Hospital in Pisa, and who were previously scheduled for a follow-up visit during the lockdown for COVID-19 (March 9, 2020-May 04, 2020) were screened for this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Glucose | One week after the end of the lockdown period
  Blood glucose was expressed in mg/dl and was determined by standard techniques.
HbA1c | One week after the end of the lockdown period
  HbA1c was expressed as percentage or mmol/l and was determined by standard techniques.
Lipid profile | One week after the end of the lockdown period
  Complete lipid profile (total cholesterol, HDL cholesterol, LDL cholesterol, Triglcerydes) were expressed in mg/dl or mmol/l and were determined by standard techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Solini, MD, PhD, Principal Investigator — University of Pisa
Locations (1):
- University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scarmozzino F, Visioli F. Covid-19 and the Subsequent Lockdown Modified Dietary Habits of Almost Half the Population in an Italian Sample. Foods. 2020 May 25;9(5):675. doi: 10.3390/foods9050675. PMID 32466106
- [Background] Bonora BM, Boscari F, Avogaro A, Bruttomesso D, Fadini GP. Glycaemic Control Among People with Type 1 Diabetes During Lockdown for the SARS-CoV-2 Outbreak in Italy. Diabetes Ther. 2020 Jun;11(6):1369-1379. doi: 10.1007/s13300-020-00829-7. Epub 2020 May 11. PMID 32395187
- [Background] Nachimuthu S, Vijayalakshmi R, Sudha M, Viswanathan V. Coping with diabetes during the COVID - 19 lockdown in India: Results of an online pilot survey. Diabetes Metab Syndr. 2020 Jul-Aug;14(4):579-582. doi: 10.1016/j.dsx.2020.04.053. Epub 2020 May 11. PMID 32416527
- [Background] Martinez-Ferran M, de la Guia-Galipienso F, Sanchis-Gomar F, Pareja-Galeano H. Metabolic Impacts of Confinement during the COVID-19 Pandemic Due to Modified Diet and Physical Activity Habits. Nutrients. 2020 May 26;12(6):1549. doi: 10.3390/nu12061549. PMID 32466598
- [Background] Di Renzo L, Gualtieri P, Pivari F, Soldati L, Attina A, Cinelli G, Leggeri C, Caparello G, Barrea L, Scerbo F, Esposito E, De Lorenzo A. Eating habits and lifestyle changes during COVID-19 lockdown: an Italian survey. J Transl Med. 2020 Jun 8;18(1):229. doi: 10.1186/s12967-020-02399-5. PMID 32513197